CLINICAL TRIAL: NCT07103551
Title: Evaluation of the Efficacy of Injectable Platelet-rich Plasma in Orthodontic Tooth Movement Acceleration With Clear Aligner Therapy
Brief Title: Evaluation of the Efficacy of Injectable Platelet-rich Plasma in Tooth Movement Acceleration With Clear Aligner
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ali Mahmoud Ali Elhewaity, Dr, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Clear Aligner and prp
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Clear Aligner Appliance
Keywords: Malocclusion; Clear aligner; Platelet-rich plasma
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clear aligner therapy only without injection of platelet-rich plasma (No Intervention): Clear aligner only without acceleration
- Clear aligner Therapy with injection of platelet-rich plasma (Experimental): Clear aligner therapy with injection of platelet-rich plasma
  Interventions: Biological: Platelet-rich plasma

INTERVENTIONS:
Biological: Platelet-rich plasma — Platelet-rich plasma used during clear aligner therapy for acceleration of Orthodontic Tooth Movement
  Arms: Clear aligner Therapy with injection of platelet-rich plasma

SUMMARY:
Aim of the study is evaluation of the efficacy of injectable platelet-rich plasma in orthodontic tooth movement acceleration with clear aligner

DETAILED DESCRIPTION:
Malocclusion is frequently viewed as detrimental to one' self-worth and overall physical, social, and mental health. On the past few years, more and more grown-up patients have persued orthodontic care and they want attractive and pleasant options instead of traditional braces. CLEAR aligners that meet this need are also subject to technological advancements in the materials used and the methods of production. Consequently, CAT has merged as the leading trend in orthodontic innovation. The primary advateges of clear aligner therapy include the option to remove while eating, enhanced oral hygiene practices, less discomfort for patients,and the capability to visualize the treatment outcome through computer applications.

Clear aligners need to be removed during eating, when drinking hot beverages that may lead to warping, while having sugary beverages, and also when cleaning teeth.

Today, numerous methods have emerged to accelerate orthodontic tooth movement, encompassing invasive,minimally invasive,and non-invasive strategies.

IN addition, the use of medications and autologous biological solutions, like platelet-rich plasma, has been suggested.

One of the recently utilized local agents to accelerate the process of orthodontic tooth movement is platelet-rich plasma.

Platelet-rich plasma is characterized as an autologous concentration of platelets within a small quantity of plasma Prepared from blood centrifuging double spin.

The application of PRP has been used in regenerative dentistry and healing acceleration in oral surgery.

PRP serves as an abundant reservoir of cytokines and contains seven essential growth factors:

* Platelet-derived growth factors .
* Transforming growth factors.
* Epidermal growth factors.
* Vascular endothelial growth factor. The diverse range of growth factors present in PRP might facilitate the simultaneous activation of both osteoblasts and osteoclasts, reinforcing the notion that PRP can influence the movement of teeth during orthodontic treatment.

Also elevated levels of cytokine production during the process of bone remodelling could accelerate tooth movement.

ELIGIBILITY:
Inclusion Criteria:

* Non-extraction cases
* Complete permanent dentition
* Good oral hygiene
* Healthy periodontal condition
* Single or double arch treatment
* No therapeutic intervention planned intermaxillary or other intraoral or extraoral appliances including lip bumper, elastics and maxillary expansion appliances
* mild to moderate crowding

Exclusion Criteria:

* Systemic medical conditions
* Dental anomalies in tooth size or shape
* Current use of anti-inflammatory medications

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Measuring the amount of tooth movement in group of clear aligner therapy and group of clear aligners with injectable platelet-rich plasma by little's irregularity index | Baseline, 3 weeks, and 6 weeks
  Little's irregularity index is used to measure the amount of tooth movement by measuring the distance between each contact points in anterior teeth before injection and after injection